CLINICAL TRIAL: NCT02987712
Title: Management of Coagulopathy in Cirrhotic Patients Undergoing Invasive Procedures: a Prospective Trial Comparing Standard Management to Thromboelastography Protocol Based Management
Brief Title: Management of Coagulopathy in Cirrhotic Patients Undergoing Invasive Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-16-IM-0703-CTIL
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Liver Cirrhosis; Coagulopathy
Keywords: Thromboelastography
MeSH Terms: conditions — Liver Cirrhosis; Hemostatic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Survey 1 (No Intervention): Common practice
- Survey 2 (Experimental): Thromboelastography based protocol
  Interventions: Other: Thromboelastography based protocol

INTERVENTIONS:
Other: Thromboelastography based protocol — patients will be treated according to a new thromboelastography based protocol
  Arms: Survey 2

SUMMARY:
Recently it has been acknowledged that cirrhotic patients present with "rebalanced hemostasis" that results from decreased levels of both pro-coagulant and anti-coagulant factors, that is not well reflected by conventional coagulation tests (CCTs). Thromboelastography (TEG) might be a more accurate tool in these patients.

Numerous guidelines on the management of the cirrhotic patient undergoing invasive procedures have been published but most of them are not evidence based. Current literature, although conflicting, is leaning towards a restrictive approach to prophylactic correction of coagulopathy when performing invasive procedures in cirrhotic patients. The investigators suspect that common practice is more liberal . Considering the well-known adverse effects of blood product administration, the aim of the study is to re-evaluate the clinical management of cirrhotic patients undergoing invasive procedures.

Study objectives: asserting whether the use of blood products prior to invasive procedures in cirrhotic coagulopathic patients can be reduced using TEG to evaluate coagulopathy in place of CCTs, evaluating the rate of complications due to blood product use, and checking how well CCT results correlate with TEG results in these patients.

This will be a prospective pre/post TEG protocol implementation study which will include two prospective surveys with a 1:1 ratio. Survey 1: prophylactic administration of FFP/PLT prior to minor invasive procedures will be based on CCTs and physicians' clinical judgement. Survey 2: management will be based on a new TEG protocol. The investigators will include cirrhotic patients with coagulopathy who are candidates for an invasive procedure. Subject will be provided with sufficient time to reach a rational, informed decision regarding participation in the study.

Data will be collected from the computer based medical record systems, the patient file and directly from the caring physician and will include a thorough medical history and conventional blood tests, including a TEG test. All subjects will be managed according to standard of care.

Primary endpoint: amount of blood product (fresh frozen plasma/platelets) units transfused in preparation for the invasive procedures.

Secondary endpoints: bleeding complications, transfusion related side effects, 90 day survival and other complications.

This will be a prospective (pre/post) study. The calculated sample size needed is 120 subjects, 60 in each group.

DETAILED DESCRIPTION:
Background

Recently there has been a change of concept regarding the hemostatic profile of patients with liver disease from "auto-anti-coagulation" to "rebalanced hemostasis". The liver synthesizes most of the factors and inhibitors of the coagulation system as well as thrombopoietin. Thus, liver disease influences the hemostatic profile both through an effect on factor/inhibitor levels and through an effect on platelet number and function. The "rebalanced hemostasis" of liver disease results from decreased levels of most proteins involved in coagulation; promotors and inhibitors. Two proteins which are elevated in this state are factor VIII and von Willebrand factor. Elevated levels of the latter compensate to some extent for the thrombocytopenia and platelet function defects. This "rebalanced" state is not well reflected by conventional coagulation tests (CCT), which are insensitive to the anticoagulant component of hemostasis. In fact, it has been shown that thrombin generation in cirrhotic patients is normal. Considering this conceptual change together with the well-known adverse effects of blood product administration the investigators seek to re-evaluate the clinical management of cirrhotic patients undergoing invasive procedures.

Thromboelastography (TEG) provides a graphic representation of clot formation and lysis. Compared with CCTs, TEG better reflects the interaction of plasma, blood cells and PLTs and better resembles the in-vivo state. Viscoelastic tests have been used for many years for coagulation monitoring and hemostatic therapy guidance during liver transplantation. Their use in hospitalized patients with liver disease has been much more limited.

Different guidelines address the issue of coagulation test abnormalities in cirrhotic patients prior to various specific invasive procedures. According to the European Association for the Study of the Liver clinical practice guidelines, in cirrhosis, hemorrhagic complications after large volume paracentesis (LVP) are infrequent and there is no data to support pre-procedural use of fresh frozen plasma (FFP) or PLTs. The authors do note that often these products are given in case of severe coagulopathy and/or thrombocytopenia, and that caution should still be exercised in patients with severe coagulopathy, and LVP avoided in the presence of disseminated intravascular coagulation. The American Association for the Study of Liver Diseases practice guidelines state that because bleeding is uncommon, routine administration of FFP or PLTs prior to paracentesis is not recommended.

Very few randomized, double-blind controlled clinical trials regarding the management of coagulation issues in patients with liver disease exist. Some guidelines note that INR should not be used alone to assess bleeding risk, that a PLT count greater than 50-60x10^9/L should be achieved prior to high-risk procedures, and that TEG may be helpful in targeting transfusion practice. Pertaining to esophageal varices, few data support the notion that coagulopathy is directly related to bleeding risk, and despite the existence of various specific guidelines on management of esophageal varices, specific recommendations on coagulation parameters for prophylactic esophageal variceal band ligation (EVBL) are missing. When prophylactic EVBL is deemed unsafe due to a coagulation disorder, they recommend avoiding it. Although it is uncertain what the optimal platelet counts should be in this situation, they recommend levels exceeding 56x10^9/L and possibly a fibrinogen level above 100-150 mg/dL. They note that FFP transfusion is problematic because of the large volume needed to "correct" the INR.

Consensus guidelines for peri-procedural management of coagulation status and hemostasis risk in percutaneous image-guided interventions conclude that central venous catheterization (CVC) can be performed safely by experienced physicians in the presence of abnormal coagulation parameters. According to an editorial in Chest, CVC insertion, even under ultrasound guidance, carries a significant risk of mechanical complications, some of which could be life threatening. The editorial states that reversal of severe thrombocytopenia or factor deficiencies may decrease the risk of bleeding in patients with severe coagulopathies, and that according to the published data, the risk-to-benefit ratio favors reversal of severe coagulopathies (e.g., PLTs 50x10^9/L and/or INR 1.5, and/or PTT 50 s). It is of note that the two aforementioned articles refer to coagulopathies as a whole and not specifically the coagulopathy of liver disease. Another study assessed the safety of CVC insertion under ultrasound guidance and the incidence of complications in patients with liver disease coagulopathy. It concluded that the incidence of major vascular and non-vascular complications was low even in the absence of prophylactic correction of coagulopathy and that the incidence of minor vascular complications was higher but acceptable and easily manageable.

A different study states that coagulopathy in cirrhotic patients undergoing surgery is a major concern for surgeons. Nonetheless, thrombocytopenia that is not severe, should not be automatically considered an index of increased bleeding risk. They state that compared with CCTs, TEG provides a better assessment of the degree of coagulopathy and offers information that can assist in managing these patients. Additionally, preoperative administration of FFP to correct the INR should be avoided due to ineffectiveness and associated complications.

There are also general guidelines for cirrhotic patients about to undergo invasive procedures, and among them guidelines regarding hemostatic management in this patient population. These apply to three clinical phases:

1. Pre-procedural phase - no prophylactic correction of hemostasis should be applied, infections should be treated and renal status optimized.
2. Intra-procedural phase - active bleeding is treated using transfusion or antifibrinolytics, a low central venous pressure (CVP) should be maintained and normal body temperature, calcium and pH should be maintained.
3. Post-procedural phase - CVP should be restored to normal and thrombotic or bleeding complications should be sought and treated.

The University of Texas Southwestern Medical Center at Dallas recently developed multidisciplinary guidelines for periprocedural transfusion of blood components in cirrhotic patients undergoing gastrointestinal procedures. For procedures with mild to moderate-risk they recommend not transfusing PLTs with counts>30x10^9/L. As for high-risk procedures, they state that PLTs may be required during the procedure with a count<30x10^9/L. They recommend transfusion of FFP only when the INR is≥2.6. Notably, a randomized controlled trial performed by De Pietry et al. evaluated TEG-guided blood product use before invasive procedures in cirrhosis with severe coagulopathy. It concluded that in patients with a significant coagulopathy before the procedure, a TEG guided infusion strategy led to a significantly lower use of blood products compared to CCT, without an increase in bleeding complications.

Finally, several publications address coagulopathy management in liver transplantation. These publications demonstrate that the method of coagulation monitoring used effects transfusion practice and that viscoelastic tests can reduce overall transfusion requirements.

Thus, it seems that the ability of CCTs to predict bleeding diathesis in cirrhotic patients is diminished, whereas TEG might be a more accurate tool. It is important to bear in mind the adverse implications of the liberal use of blood products. It seems that the current literature, although conflicting, is leaning towards a more restrictive approach to prophylactic correction of coagulopathy when performing invasive procedures in cirrhotic patients. Based on the literature and on clinical experience, the investigators suspect that common practice is more liberal and that in practice prophylactic correction of coagulation laboratory tests abnormalities is more common than it should be based on published guidelines.

Objectives

* Assert whether the use of blood products prior to invasive procedures in cirrhotic coagulopathic patients can be reduced using TEG to evaluate coagulopathy in place of CCTs.
* Evaluate the rate of complications due to blood product use in these patients.
* Check the correlation between CCT results and TEG in these patients.

Methods and Materials

Study Design

This will be a prospective pre/post TEG protocol implementation study. It will include two prospective surveys with a 1:1 ratio. A full and thorough medical history will be obtained. Medical conditions, past surgeries, medications currently in use and laboratory test results (including TEG) will be noted. In addition, the type of procedure the patient is undergoing will be recorded along with bleeding complications, blood product transfusion record, transfusion related side effects and complications, any other complication that can be attributed the procedure or to its avoidance, total hospital stay from the time of the procedure until hospital release and 90-day survival following the procedure.

Subjects will be consecutively enrolled, in accordance with selection criteria in the two surveys:

1. Survey 1 - will be performed at baseline. Management will be based on CCTs, as per common practice.
2. Survey 2 - management will be based on the TEG result. According to the new TEG protocol, subjects with a reaction time (r)>12 min will receive FFP, and patients with a maximum amplitude (MA)<36 mm will receive PLTs.

All subjects will be managed according to standard of care.

Regulatory Requirements

This study protocol complies with the declaration of Helsinki and will be conducted according to rules and guidelines of good clinical practice (GCP).

Informed Consent

Informed consent will be obtained from the subjects by an authorized research team member only. Subject will be provided with sufficient time to reach a rational, informed decision regarding participation in the study.

Subject Confidentiality

Access to data will be granted to authorized study members only. The Case Report Form (CRF) will contain patient identification number. Any subjects' personal information will be removed from the CRF after the completion of the form and its integration to the database.

Sample Size

The study will include a total of 120 subjects, 60 in each group, in order to compensate for dropouts. Sample size was calculated using the WINPEPI program. Version 11.24.

Statistical Analysis

the investigators intend to assess the influence of the use of a TEG related protocol on the use of blood products in cirrhotic patients. They will examine the relationship of each of the factors predicting blood product use and demographic data to use of blood product. Quantitative data with normal distribution will be evaluated using t-test for independent samples. In case the assumptions for parametric tests will not hold true, quantitative data will be evaluated using an a-parametric Mann-Whitney test. Continuous data will be presented as average±SD. Dichotomous data will be evaluated using the chi-square test. Fisher exact test will be used when more than 20% of the expected observations were less than 5 or any expected observation was less than 2. Categorical data will be presented as a number of cases and percent. Multivariate logistic regression analysis will be used for the primary outcome and exposure (blood product use prevalence and predicting and demographic factors) in order to determine independent risk factors. The data included in the multivariate logistic regression model will be significant demographic data and data found to have a Pv<0.1 in the univariate analysis. A Pv of 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Follow up at the Gastroenterology Unit at TLVMC
* Diagnosis of cirrhosis
* Abnormal coagulation test results: INR > 1.5 and/or a PLT count < 50x10^9/L
* Planned to undergo an invasive procedure
* Hospitalization in one of the following units at TLVMC: Internal Medicine D, Internal Medicine T, Internal Medicine Consultations, Intensive Care Unit, Surgical Intensive Care Unit, General Surgery Division and the Gastroenterology unit.
* Invasive procedures: central venous catheter placement, drainage of ascitic fluid, endoscopic procedures (variceal ligation or polypectomy) or any surgical procedure (excluding liver transplantation).

Exclusion Criteria:

* Ongoing bleeding
* Current/recent (past 7 days) antiplatelet/anticoagulant therapy
* Hemodialysis in the previous 7 days.
* planned procedure is liver transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Amount of blood product (FFP/PLT) units transfused in preparation for the invasive procedures. | Intraoperative
  Number of FFP/PLT units transfused

SECONDARY OUTCOMES:
Bleeding complications. | up to 30 days from procedure performance or death, whichever comes first
  Number of episodes of overt bleeding / hemoglobin drop requiring transfusion
Transfusion-related side effects | up to 30 days from procedure performance or death, whichever comes first
  Number and type of side effects attributable to blood product administration
90-day survival | Up to 90 days from procedure performance
Other complications | up to 30 days from procedure performance or death, whichever comes first
  Number and type of complication that can be attributed the procedure or to avoidance of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Idit Matot, MD, PhD, Principal Investigator — Tel-Aviv Sourasky Medical Center

IPD SHARING:
Plan to Share IPD: No
we do not plan to share IPD

REFERENCES:
- [Background] Weeder PD, Porte RJ, Lisman T. Hemostasis in liver disease: implications of new concepts for perioperative management. Transfus Med Rev. 2014 Jul;28(3):107-13. doi: 10.1016/j.tmrv.2014.03.002. Epub 2014 Mar 15. PMID 24721432
- [Background] Tripodi A, Mannucci PM. The coagulopathy of chronic liver disease. N Engl J Med. 2011 Jul 14;365(2):147-56. doi: 10.1056/NEJMra1011170. No abstract available. PMID 21751907
- [Background] Tripodi A, Salerno F, Chantarangkul V, Clerici M, Cazzaniga M, Primignani M, Mannuccio Mannucci P. Evidence of normal thrombin generation in cirrhosis despite abnormal conventional coagulation tests. Hepatology. 2005 Mar;41(3):553-8. doi: 10.1002/hep.20569. PMID 15726661
- [Background] Salooja N, Perry DJ. Thrombelastography. Blood Coagul Fibrinolysis. 2001 Jul;12(5):327-37. doi: 10.1097/00001721-200107000-00001. PMID 11505075
- [Background] Mallett SV, Chowdary P, Burroughs AK. Clinical utility of viscoelastic tests of coagulation in patients with liver disease. Liver Int. 2013 Aug;33(7):961-74. doi: 10.1111/liv.12158. Epub 2013 May 3. PMID 23638693
- [Background] European Association for the Study of the Liver. EASL clinical practice guidelines on the management of ascites, spontaneous bacterial peritonitis, and hepatorenal syndrome in cirrhosis. J Hepatol. 2010 Sep;53(3):397-417. doi: 10.1016/j.jhep.2010.05.004. Epub 2010 Jun 1. No abstract available. PMID 20633946
- [Background] Runyon BA; AASLD Practice Guidelines Committee. Management of adult patients with ascites due to cirrhosis: an update. Hepatology. 2009 Jun;49(6):2087-107. doi: 10.1002/hep.22853. No abstract available. PMID 19475696
- [Background] Northup PG, Caldwell SH. Coagulation in liver disease: a guide for the clinician. Clin Gastroenterol Hepatol. 2013 Sep;11(9):1064-74. doi: 10.1016/j.cgh.2013.02.026. Epub 2013 Mar 16. PMID 23506859
- [Background] Patel IJ, Davidson JC, Nikolic B, Salazar GM, Schwartzberg MS, Walker TG, Saad WA; Standards of Practice Committee, with Cardiovascular and Interventional Radiological Society of Europe (CIRSE) Endorsement. Consensus guidelines for periprocedural management of coagulation status and hemostasis risk in percutaneous image-guided interventions. J Vasc Interv Radiol. 2012 Jun;23(6):727-36. doi: 10.1016/j.jvir.2012.02.012. Epub 2012 Apr 17. No abstract available. PMID 22513394
- [Background] Baron RM. Point: should coagulopathy be repaired prior to central venous line insertion? Yes: why take chances? Chest. 2012 May;141(5):1139-1142. doi: 10.1378/chest.11-3225. No abstract available. PMID 22553259
- [Background] Singh SA, Sharma S, Singh A, Singh AK, Sharma U, Bhadoria AS. The safety of ultrasound guided central venous cannulation in patients with liver disease. Saudi J Anaesth. 2015 Apr-Jun;9(2):155-60. doi: 10.4103/1658-354X.152842. PMID 25829903
- [Background] Lopez-Delgado JC, Ballus J, Esteve F, Betancur-Zambrano NL, Corral-Velez V, Manez R, Betbese AJ, Roncal JA, Javierre C. Outcomes of abdominal surgery in patients with liver cirrhosis. World J Gastroenterol. 2016 Mar 7;22(9):2657-67. doi: 10.3748/wjg.v22.i9.2657. PMID 26973406
- [Background] Yates SG, Gavva C, Agrawal D, Sarode R. How do we transfuse blood components in cirrhotic patients undergoing gastrointestinal procedures? Transfusion. 2016 Apr;56(4):791-8. doi: 10.1111/trf.13495. Epub 2016 Feb 15. PMID 26876945
- [Background] De Pietri L, Bianchini M, Montalti R, De Maria N, Di Maira T, Begliomini B, Gerunda GE, di Benedetto F, Garcia-Tsao G, Villa E. Thrombelastography-guided blood product use before invasive procedures in cirrhosis with severe coagulopathy: A randomized, controlled trial. Hepatology. 2016 Feb;63(2):566-73. doi: 10.1002/hep.28148. Epub 2015 Dec 9. PMID 26340411
- [Background] Coakley M, Reddy K, Mackie I, Mallett S. Transfusion triggers in orthotopic liver transplantation: a comparison of the thromboelastometry analyzer, the thromboelastogram, and conventional coagulation tests. J Cardiothorac Vasc Anesth. 2006 Aug;20(4):548-53. doi: 10.1053/j.jvca.2006.01.016. Epub 2006 Apr 19. PMID 16884987
- [Background] Wang SC, Shieh JF, Chang KY, Chu YC, Liu CS, Loong CC, Chan KH, Mandell S, Tsou MY. Thromboelastography-guided transfusion decreases intraoperative blood transfusion during orthotopic liver transplantation: randomized clinical trial. Transplant Proc. 2010 Sep;42(7):2590-3. doi: 10.1016/j.transproceed.2010.05.144. PMID 20832550